CLINICAL TRIAL: NCT00820755
Title: Open, Randomized, Multinational Phase IIIb Trial Evaluating the Activity and Safety of Cetuximab as 250 mg/m^2 Weekly and 500 mg/m^2 Every Two Weeks Maintenance Therapy After Platinum-based Chemotherapy in Combination With Cetuximab as First-line Treatment for Subjects With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Trial With Cetuximab in Maintenance Therapy After Platinum Based Chemotherapy in First Line Treatment of Non-small Cell Lung Cancer (NSCLC)
Acronym: NEXT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62240-506
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

ARMS (3):
- Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy (Active Comparator)
  Interventions: Drug: Cetuximab plus Platinum-based Doublet Chemotherapy
- Cetuximab 500 mg/m^2 every 2 weeks (Active Comparator)
  Interventions: Drug: Cetuximab 500 mg/m^2
- Cetuximab 250 mg/m^2 weekly (Active Comparator)
  Interventions: Drug: Cetuximab 250 mg/m^2

INTERVENTIONS:
Drug: Cetuximab plus Platinum-based Doublet Chemotherapy — Single first dose of cetuximab 400 mg/m^2 infusion will be administered intravenously over 120 minutes (min) followed by cetuximab 250 mg/m^2 intravenous infusion over 60 min q1w with background platinum-based doublet chemotherapy up to maximum of 6 cycles, until progressive disease, unacceptable toxicity, or withdrawal of consent. Platinum based doublet chemotherapy will be administered as intravenous infusion as per study center included: vinorelbine 25 mg/m^2 on Day 1 (D1) and Day 8 (D8)+cisplatin 80 mg/m^2 on D1; or gemcitabine 1250 mg/m^2 on D1 and D8+cisplatin 75 mg/m^2 on D1; or gemcitabine 1000 mg/m^2 on D1 and D8+carboplatin at dose to reach area under curve (AUC)5 milligram*hour/milliliter (mg*hr/mL) on D1; or Docetaxel 75 mg/m^2 on D1+cisplatin 75 mg/m^2 on D1; or paclitaxel 175 mg/m^2 on D1+cisplatin 80 mg/m^2 on D1; or paclitaxel 200 mg/m^2 on D1+carboplatin at dose to reach AUC6 mg*hr/mL on D1, of each 3-week treatment cycle for a maximum of 6 cycles.
  Arms: Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy
Drug: Cetuximab 500 mg/m^2 — Subjects who will be free of disease progression at the end of combination therapy, will enter in the maintenance therapy period. In the maintenance period, subjects will be receive cetuximab 500 mg/m^2 as intravenous infusion every 2 weeks, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
  Other Names: Erbitux
  Arms: Cetuximab 500 mg/m^2 every 2 weeks
Drug: Cetuximab 250 mg/m^2 — Subjects who will free of disease progression at the end of combination therapy, will enter in the maintenance therapy period. In the maintenance period, subjects will be receive cetuximab 250 mg/m^2 as intravenous infusion weekly, until PD, unacceptable toxicity, or withdrawal of consent.
  Other Names: Erbitux
  Arms: Cetuximab 250 mg/m^2 weekly

SUMMARY:
This open-label, randomized, multinational, non-comparative, phase IIIb trial with 2 parallel groups will screen about 1400 subjects with stage IIIB non-small cell lung cancer (NSCLC) with pleural effusion or stage IV NSCLC. It is expected that of approximately 1200 (85 percent) subjects who will be included, about 1000 will be Caucasian; about 120 Asian, and the remainder (about 80) will be of other ethnic origin (that is neither Caucasian nor Asian). Approximately 480 (40 percent) subjects are expected to be free of progression at the end of combination treatment with cetuximab and platinum-based chemotherapy. These subjects will be eligible for randomization to intravenous cetuximab maintenance therapy with either 500 milligram per square meter (mg/m^2) every 2 weeks or 250 mg/m^2 weekly (q1w); about 240 subjects are expected per group.

The trial will be performed in a community practice setting, with approximately 230 centers participating in the trial worldwide (planned countries are Argentina, Australia, Austria, Belgium, Brazil, Chile, China, Colombia, Czech Republic, France, Germany, Greece, Hong Kong, Hungary, India, Ireland, Israel, Italy, Mexico, Netherlands, Poland, Portugal, Russia, Singapore, Slovakia, South Africa, South Korea, Spain, Switzerland, Taiwan, Turkey, United Kingdom and Venezuela). With noncompetitive enrollment, approximately 4 to 8 subjects are expected to be enrolled at each center. Enrollment in the individual centers is generally limited to a maximum of 8 subjects. If any of these subjects does not receive trial treatment for any reason or discontinue all trial treatment at the first visit, additional subjects may be enrolled until 8 subjects were treated. The primary endpoint of the trial will be overall survival time from inclusion into the trial to death. Additional secondary efficacy endpoints will be time to treatment failure, tumor response, and disease control rate. Other endpoints will include safety and toxicity, compliance with maintenance therapy, subject satisfaction and translational research (TR) (for subjects with tumor samples available).

ELIGIBILITY:
Inclusion Criteria:

* Subject has given written informed consent before any trial-related activities are carried out
* Male or female, greater than or equal to (>=)18 years of age at the time of informed consent, inpatient or outpatient
* Diagnosis of histologically or cytologically confirmed NSCLC, stage IIIB NSCLC with pleural effusion or stage IV
* Presence of at least 1 uni-dimensionally measurable index lesion, whereby index lesions must not lie in a previously irradiated area
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at inclusion in the trial
* White blood count>= 3 * 10^9 per liter (/L) with neutrophils >= 1.5 * 10^9 /L , platelet count >=100 * 10^9 /L , and hemoglobin >= 5.6 millimole per liter (mmol/L) (9 gram per deciliter [g/dL])
* Total bilirubin less than or equal to (=<)1.5 * upper limit of normal (ULN) range
* Aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) =< 5 * ULN
* Glomerular filtration rate (GFR) >=60 milliliter per minute (mL/min). The creatinine clearance (CrCl) estimated based on the Cockroft-Gault formula is used as a surrogate for the GFR
* Effective contraception that is, barrier method (condoms, diaphragm), oral, injectable or implant birth control, for both male and female subjects during the whole trial period and for at least 6 months after the end of trial treatment, if the risk of conception exists
* Recovered from relevant toxicities prior to inclusion in the trial

Exclusion Criteria:

* Previous exposure to Epidermal Growth Factor Receptor (EGFR)-targeting therapy
* Previous chemotherapy for NSCLC; neo-adjuvant or adjuvant (radio-)chemotherapy is allowed if it was finished 6 months prior to start of trial treatment
* Major surgery within 30 days prior to inclusion in the trial
* Prior chest irradiation within 90 days prior to inclusion in the trial (palliative radiation of bone lesions is allowed)
* Participation in another clinical trial or treatment with any investigational agent(s) within 30 days prior to inclusion in the trial
* Concurrent chronic systemic immune therapy, chemotherapy for disease other than cancer, or hormone therapy for the treatment of cancer not indicated in the trial protocol
* Documented or symptomatic brain metastasis
* Pre-existing ascites Grade >= 2 and/or pericardial effusion Grade >= 2
* Superior vena cava syndrome contra-indicating hydration
* Previous malignancy in the last 5 years except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Active infection (infection requiring intravenous antibiotics), including active tuberculosis, known and declared human immunodeficiency virus (HIV)
* Myocardial infarction within 6 months prior to inclusion into the trial, uncontrolled congestive heart failure; or any current Grade 3 or 4 cardio-vascular disorder despite treatment
* Known hypersensitivity reaction to any of the components of trial treatments
* Symptomatic peripheral neuropathy National Cancer Institute-Common Toxicity Criteria (NCI-CTC) Grade >= 2 and/or ototoxicity Grade >= 2, except if due to trauma or mechanical impairment due to tumor mass
* History of significant neurologic or psychiatric disorders including dementia, seizures, bipolar disorder
* Medical or psychological condition that would not permit the subject to complete the trial or sign informed consent
* Legal incapacity or limited legal capacity
* Known drug abuse
* Pregnancy (absence to be confirmed by serum beta-human chorionic gonadotropin [beta-HCG test]) or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Heeger, MD MSc, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Central Contact, Darmstadt, Germany

REFERENCES:
- [Derived] Heigener DF, Pereira JR, Felip E, Mazal J, Manzyuk L, Tan EH, Merimsky O, Sarholz B, Esser R, Gatzemeier U. Weekly and every 2 weeks cetuximab maintenance therapy after platinum-based chemotherapy plus cetuximab as first-line treatment for non-small cell lung cancer: randomized non-comparative phase IIIb NEXT trial. Target Oncol. 2015 Jun;10(2):255-65. doi: 10.1007/s11523-014-0336-7. Epub 2014 Sep 9. PMID 25195590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participants (informed consent): January 2009/17 March 2010. Clinical data cut-off: 17 December 2011
Pre-assignment Details: Enrolled: 673 screened for eligibility; 90 excluded (mainly non-fulfillment of inclusion or exclusion criteria). 583 participants started.
Groups:
- Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy: Combination Phase: Single first dose of cetuximab 400 milligram per square meter (mg/m^2) infusion administered intravenously over 120 minutes (min) followed by cetuximab 250 mg/m^2 intravenous infusion over 60 min weekly (q1w) with background platinum-based doublet chemotherapy up to maximum of 6 cycles, until progressive disease, unacceptable toxicity, or withdrawal of consent. Platinum based doublet chemotherapy infusion intravenously as per study center included: vinorelbine 25 mg/m^2 on Day 1 (D1) and Day 8 (D8)+cisplatin 80 mg/m^2 on D1; or gemcitabine 1250 mg/m^2 on D1 and D8+cisplatin 75 mg/m^2 on D1; or gemcitabine 1000 mg/m^2 on D1 and D8+carboplatin at dose to reach area under curve (AUC)5 mg*hour/milliliter (mg*h/mL) on D1; or Docetaxel 75 mg/m^2 on D1+cisplatin 75 mg/m^2 on D1; or paclitaxel 175 mg/m^2 on D1+cisplatin 80 mg/m^2 on D1; or paclitaxel 200 mg/m^2 on D1+carboplatin at dose to reach AUC6 mg*h/mL on D1, of each 3-week treatment cycle for a maximum of 6 cycles.
- Cetuximab 500 mg/m^2 Every 2 Weeks: Participants who were free of disease progression at the end of combination therapy, entered in the maintenance therapy period. In the maintenance period, participants received cetuximab 500 mg/m^2 as intravenous infusion every 2 weeks, until progressive disease (PD), unacceptable toxicity, or withdrawal of consent.
- Cetuximab 250 mg/m^2 Weekly: Participants who were free of disease progression at the end of combination therapy, entered in the maintenance therapy period. In the maintenance period, participants received cetuximab 250 mg/m^2 as intravenous infusion weekly, until PD, unacceptable toxicity, or withdrawal of consent.
Period: Period 1: Combination Therapy Phase
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Started | 583 | 0 | 0
Completed | 313 (2 of 313 participants excluded from maintenance phase analysis (reason: not eligible)) | 0 | 0
Not Completed | 270 | 0 | 0
Not completed — Adverse Event | 77 | 0 | 0
Not completed — Death | 28 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0
Not completed — Progressive disease | 114 | 0 | 0
Not completed — Sympt. deterioration w/o PD by imaging | 14 | 0 | 0
Not completed — Other | 11 | 0 | 0
Period: Period 2: Maintenance Therapy Phase
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Started | 0 | 157 | 154
Completed | 0 | 112 | 109
Not Completed | 0 | 45 | 45
Not completed — Investigational study phase ongoing | 0 | 45 | 45

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy
Number analyzed (Participants) | 583
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147
  Male | 436

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: The OS time is defined as the time from trial inclusion to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whichever is earlier.
Time Frame: Time from trial inclusion to death or last day known to be alive, reported between day of first participant included, that is, Jan 2009 until cut-off date (17 Dec 2011)
Population: Intention-to-treat (ITT) maintenance analysis set included all participants who were included in ITT (all the participants enrolled in this study) analysis set, judged to be progression-free (based on computer tomography [CT] or magnetic resonance imaging [MRI] scan) by the Investigator and randomized to maintenance therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
months | 16.1 [13.6 to 18.2] | 15.5 [13.2 to 19.7]

2. Secondary Outcome: Overall Survival (OS) Time (From Randomization to Cetuximab Maintenance Regimen Until Death)
Description: The OS time is defined as the time from randomization in cetuximab maintenance regimen to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whichever is earlier.
Time Frame: Time from randomization in cetuximab maintenance regimen to death or last day known to be alive, reported between day of first participant randomized, that is, May 2009 until cut-off date (17 Dec 2011)
Population: ITT maintenance analysis set included all participants who were included in ITT (all the participants enrolled in this study) analysis set, judged to be progression-free (based on CT or MRI scan) by the Investigator and randomized to maintenance therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
months | 12.6 [10.1 to 14.8] | 12.6 [9.3 to 16.0]
Statistical Analysis 1: Comparison: Cetuximab 500 mg/m^2 Every 2 Weeks vs Cetuximab 250 mg/m^2 Weekly; Exploratory analysis to test the null hypothesis of no difference between maintenance therapy regimen. Model is adjusted by histology (interactive voice response system [IVRS]) and tumor response status at the end of combination therapy ('complete response [CR] or partial response [PR]' versus 'other'); Test type: Superiority or Other; p = 0.1265, Log Rank; Hazard Ratio, log = 0.959, 95% CI 2-sided [0.736 to 1.250]

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from trial inclusion to date of either first occurrence of progression, discontinuation of treatment due to progression or adverse event, withdrawal of consent or lost to follow up, start of further anticancer therapy, or death, whichever is earlier. Participants without events are censored either at the time of their last drug intake, or on the day of inclusion (Day 1) if they received no study drug.
Time Frame: Time from trial inclusion to treatment failure or last drug intake, reported between day of first participant included, that is, Jan 2009 until cut-off date (17 Dec 2011)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
months | 5.8 [5.6 to 6.6] | 6.6 [6.1 to 6.9]

4. Secondary Outcome: Time to Treatment Failure (From Randomization to Cetuximab Maintenance Regimen Until Death)
Description: Time from randomization in cetuximab maintenance regimen to date of either first occurrence of progression, discontinuation of treatment due to progression or adverse event, withdrawal of consent or lost to follow up, start of further anticancer therapy, or death, whichever is earlier. Participants without events are censored either at the time of their last drug intake, or on the day of randomization (Day 1 of maintenance therapy) if they received no study drug.
Time Frame: Time from randomization in cetuximab maintenance regimen to treatment failure or last drug intake, reported between day of first participant randomized, that is, May 2009 until cut-off date (17 Dec 2011)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
months | 2.6 [2.1 to 2.8] | 2.8 [2.6 to 4.0]
Statistical Analysis 1: Comparison: Cetuximab 500 mg/m^2 Every 2 Weeks vs Cetuximab 250 mg/m^2 Weekly; Exploratory analysis to test the null hypothesis of no difference between maintenance therapy regimen. Model is adjusted by histology (IVRS) and tumor response status at the end of combination therapy ('CR or PR' versus 'other'); Test type: Superiority or Other; p = 0.0622, Log Rank; Hazard Ratio (HR) = 0.774, 95% CI [0.613 to 0.976]

5. Secondary Outcome: Percentage of Participants With Best Unconfirmed Tumor Response in the Combination Therapy Phase
Description: The response rate is defined as the percentage of participants having achieved complete response (CR) or partial response (PR) as the unconfirmed best overall response (BOR) according to centrally reviewed investigator assessments based on an independent review charter (IRC). As per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: CR = Disappearance of all target lesions; PR = at least 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Evaluations were performed every 2 cycles during combination therapy period until progression and at the end of combination therapy period, reported between day of first participant included, that is, Jan 2009, until cut-off date, (17 Dec 2011)
Population: ITT analysis set included all participants enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy
Number analyzed (Participants) | 583
percentage of participants | 36.2 [32.3 to 40.2]

6. Secondary Outcome: Percentage of Participant With Best Unconfirmed Tumor Response for the Whole Study Period
Description: The response rate is defined as the percentage of participants having achieved CR and PR as the BOR according to IRC assessment in combination therapy phase and radiological assessments (based on response evaluation criteria in solid tumors [RECIST] Version 1.0) in the maintenance therapy phase. As per RECIST v1.0 for target lesions and assessed by MRI: CR = Disappearance of all target lesions; PR = at least 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Evaluations were performed every 2 cycles during combination therapy and 6-weekly during maintenance therapy period until progression and at end of both periods, reported between day of first participant included, Jan 2009 until cut-off date (17 Dec 2011)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
percentage of participants | 54.8 [46.6 to 62.7] | 57.8 [49.6 to 65.7]

7. Secondary Outcome: Percentage of Participants With Disease Control in the Combination Therapy Phase
Description: The disease control rate is defined as the percentage of participants having achieved complete response or partial response or stable disease as the unconfirmed BOR according to IRC assessment.
Time Frame: as for outcome 5
Population: ITT analysis set included all participants enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy
Number analyzed (Participants) | 583
percentage of participants | 65.7 [61.7 to 69.5]

8. Secondary Outcome: Percentage of Participants With Disease Control for the Whole Study Period
Description: The disease control rate is defined as the percentage of participants having achieved complete response or partial response or stable disease as the unconfirmed best overall response according to IRC assessment in combination therapy phase and radiological assessments (based on RECIST Version 1.0 criteria) in the maintenance therapy phase.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
percentage of participants | 98.7 [95.5 to 99.8] | 99.4 [96.4 to 100]

9. Primary Outcome: Percentage of Participants With 1-year Overall Survival
Description: The OS time is defined as the time from trial inclusion to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whichever is earlier. Percentage of participants who were still alive until one year after the last participant was included (March 2010).
Time Frame: Time from trial inclusion to death or last day known to be alive, reported between day of first participant included, that is, Jan 2009 until one year after the last participant was included (March 2010)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Number analyzed (Participants) | 157 | 154
percentage of participants | 62.8 [54.7 to 70.0] | 64.4 [56.2 to 71.4]

ADVERSE EVENTS:
Time Frame: Time from Baseline up to 30 days after the last dose of study treatment.
Description: One participant who was randomized to 'Cetuximab 500 mg/m^2 Every 2 Weeks' arm actually received 'Cetuximab 250 mg/m^2 Weekly' treatment and was counted in this group for safety analysis
Groups:
- Cetuximab 500 mg/m^2 Every 2 Weeks: Participants who were free of disease progression after combination therapy, they administered with cetuximab 500 mg/m^2 intravenously for 2 weeks, for up to PD, development of unacceptable toxicities, or withdrawal of consent after the end of combination therapy.
Arm/Group | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy | Cetuximab 500 mg/m^2 Every 2 Weeks | Cetuximab 250 mg/m^2 Weekly
Serious Adverse Events (participants affected / at risk) | 243/583 | 30/156 | 33/155
Other Adverse Events (participants affected / at risk) | 564/583 | 121/156 | 136/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy (N=583) | Cetuximab 500 mg/m^2 Every 2 Weeks (N=156) | Cetuximab 250 mg/m^2 Weekly (N=155)
Anaemia (Blood and lymphatic system disorders) | 6 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 8 | 1 | 0
Fatigue (General disorders) | 6 | 0 | 1
Pyrexia (General disorders) | 9 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Platelet count decreased (Investigations) | 5 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 0
Febdrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 20 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 32 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Arrhythmia superaventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 1
Electromechanical dissociation (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 3 | 2 | 0
Device leakage (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 2 | 2 | 1
General physical health deterioration (General disorders) | 4 | 1 | 0
Infusion related reaction (General disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 2 | 0 | 0
Organ failure (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 3 | 0 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 8 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 0 | 0
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 17 | 4 | 4
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0
Pyothorax (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 0
C-Reactive protein increased (Investigations) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 3 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Pyramidal tract syndrome (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 1
Femoral artery embolism (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 3 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab 250 mg/m^2 q1w + Platinum-based Doublet Chemotherapy (N=583) | Cetuximab 500 mg/m^2 Every 2 Weeks (N=156) | Cetuximab 250 mg/m^2 Weekly (N=155)
Anaemia (Blood and lymphatic system disorders) | 134 | 9 | 15
Leukopenia (Blood and lymphatic system disorders) | 72 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 208 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 112 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 13 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 21 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 31 | 0 | 0
Constipation (Gastrointestinal disorders) | 109 | 3 | 12
Diarrhoea (Gastrointestinal disorders) | 120 | 6 | 15
Dyspepsia (Gastrointestinal disorders) | 36 | 0 | 0
Nausea (Gastrointestinal disorders) | 212 | 3 | 9
Odynophagia (Gastrointestinal disorders) | 5 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 47 | 0 | 0
Vomiting (Gastrointestinal disorders) | 122 | 2 | 8
Asthenia (General disorders) | 124 | 6 | 16
Chills (General disorders) | 16 | 0 | 0
Fatigue (General disorders) | 114 | 7 | 13
Influenza like illness (General disorders) | 11 | 0 | 0
Mucosal Inflammation (General disorders) | 67 | 0 | 0
Non-cardiac chest pain (General disorders) | 23 | 8 | 7
Oedema peripheral (General disorders) | 21 | 0 | 0
Pyrexia (General disorders) | 69 | 9 | 10
Paronychia (Infections and infestations) | 30 | 9 | 12
Upper respiratory tract infection (Infections and infestations) | 24 | 0 | 0
Alanine aminotransferase increased (Investigations) | 26 | 0 | 0
Haemoglobin decreased (Investigations) | 40 | 0 | 0
Neutrophil count decreased (Investigations) | 19 | 0 | 0
Platelet count decreased (Investigations) | 40 | 0 | 0
White blood cell count decreased (Investigations) | 20 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 112 | 8 | 13
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 69 | 9 | 14
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 5 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 6 | 8
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 0 | 0
Dizziness (Nervous system disorders) | 35 | 4 | 8
Dysgeusia (Nervous system disorders) | 28 | 0 | 0
Headache (Nervous system disorders) | 29 | 7 | 9
Neuropathy peripheral (Nervous system disorders) | 26 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 8 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 38 | 9 | 6
Insomnia (Psychiatric disorders) | 31 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 69 | 14 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 49 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 20 | 22
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 306 | 40 | 40
Alopecia (Skin and subcutaneous tissue disorders) | 109 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 83 | 11 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 51 | 10 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 46 | 9 | 11
Acne (Skin and subcutaneous tissue disorders) | 31 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Hypertension (Vascular disorders) | 19 | 0 | 0
Phlebitis (Vascular disorders) | 13 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 7 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 10 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 11 | 13

LIMITATIONS AND CAVEATS:
Enrollment was stopped prematurely when cetuximab did not gain regulatory approval in this indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other